CLINICAL TRIAL: NCT02514837
Title: Microwave Radiometry for the Diagnosis and Monitoring of Breast Cancer
Acronym: RTM
Status: Withdrawn | Type: Observational
Why Stopped: No funding
Sponsor: University of Edinburgh (Other)
Responsible Party: Sponsor
Other Study IDs: RTM 2015
Record Dates: First submitted 2015-07-07; First posted 2015-08-04 (Estimated); Last update posted 2022-08-19 (Actual); Status verified 2017-05

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Temperature measured by RTM device: Both the internal temperature and skin temperature will be measured non-invasively through the skin.
  Interventions: Device: RTM

INTERVENTIONS:
Device: RTM — Both the internal temperature and skin temperature will be measured non-invasively through the skin using the RTM device

SUMMARY:
A malignant tumor has higher temperature than normal tissue and the temperature of the tumor is dependent on the tumor growth rate. Thus tumor temperature is the universal indicator of tumor activity.

The temperature changes begin in the stage of atypical hyperplasia and increased proliferation and this opens up the possibilities for detection of patients with high risk lesions.

Microwave radiometer (RTM-01-RES) allows measurement of temperature changes of internal tissue at the depth of several centimetre and allows visualization of the temperature on the thermogram and temperature field.

It is noninvasive and the measurement of internal temperature is based on receiving natural electromagnetic radiation from the tissue in the gigahertz (GHz) frequency range. The device is absolutely harmless and has no risk because it does not emit any radiation. It can be used repeatedly as a method of monitoring.

Microwave radiometry has successfully completed seven clinical trials of more than 1000 patients in different countries. Microwave device (RTM-01-RES) is used in more than 300 medical centers in 30 countries.

Medical technology of microwave radiometry is included in the nomenclature of medical services in the Russian Federation, the Ministry of Health and is part of the standard of care for patients with malignant tumors of the breast.

This method of microwave radiometry is recommended by leading Russian mammalogists in the National guidelines of breast care.

The investigators would like to use the device in clinics in Scotland and later United Kingdom (UK) for breast diagnosis and monitoring treatment.

During 3 months the investigators aim to examine 150 patients with breast cancer and 150 patients without cancer who will be the control group. The results of temperature measurement will be compared with the results of histology, in particular, tumour cellulants p53 expression and other gene expression data for metabolic biomarkers and other tumor indicator. Statistical analysis of data will be performed. The device and initial training will be provided by RES Company (device producer).

DETAILED DESCRIPTION:
The temperature of a malignant tumour is a universal indicator of the growth rate of the tumor.

Tumor temperature can be used as a prediction of the benefit of individual therapies and in monitoring the efficacy of breast cancer treatment.

The temperature of tissue around a malignant tumour is correlated with micro vessel density (MVD) - the main indicator of angiogenesis.

A traditional infrared camera allows measurement of the temperature of the skin and the breast tumor at a depth of several centimetres.

It is well known that it is possible to detect thermal abnormality of internal tissues with the help of measuring the natural electromagnetic radiation in microwave frequency range. Microwave radiometer (RTM-01-RES) allows one to measure noninvasively any temperature changes of internal tissue at the depth of several centimetres and visualize the internal temperature on the thermogram and temperature field.

It was shown that the device can be used for detection of carotid temperature abnormalities and the temperature of the carotid is a good correlation to the risk of stroke in the patient.

Today it is technically possible to obtain non-invasively the information concerning thermal activity of the tumor and use this information for the prediction of individual therapies and monitoring the efficacy of breast cancer treatment.

The clinical trials in Russia show that tumors with a low degree of malignancy have low temperature changes and the tumor with high degree of malignancy have high temperature changes.

Seven clinical trials of (RTM-01-RES) with 1000 patients have shown that 90% of breast malignant tumours have substantial temperature changes (the sensitivity is 85%-95%, specificity 56%-75%).

The standard of care for patients with malignant tumors of the breast is to use microwave radiometry and this is recommended by leading Russian mammalogists in the National guidelines of breast care.

Given that the temperature of a malignant tumor is higher than a benign lesion and that the temperature of more proliferative and thus poorer outlook cancers is greater than less proliferative cancers, the aim is whether with the most up to date technology these temperatures can be measured accurately on the skin.

The benefits of such a device would be

1. Diagnostic - to help differentiate benign from malignant lesions.
2. Prognostic - to provide insight into the proliferation rate using a non-invasive test.
3. Predictive of benefit - to show that changes in temperature predate changes in tumors volume in patients treated with drug therapy initially.

The investigation is non-invasive. If it were possible to demonstrate benefit, then this simple non-invasive test could have a useful role in assessing patients with breast lumps and in particularly breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients attending the breast clinic undergoing mammography and/or ultrasound who can give written informed consent.
* The investigators aim to recruit 150 patients likely to have breast cancer clinically and 150 patients who have normal breasts/benign abnormalities.

Exclusion Criteria:

* Patients unable to give written informed consent.
* Patients not having appropriate imaging (mammography +/- ultrasound).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: no applicable; study withdrawn
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-09 (Estimated); Primary Completion 2020-02 (Estimated); Study Completion 2020-02 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of the RTM device | Results obtained from the RTM device will be compared with those obtained by conventional diagnostic techniques at 6 months.

SECONDARY OUTCOMES:
Predictability of the method | Results obtained from the RTM device will be compared with those obtained by conventional diagnostic techniques at 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Dixon, MD, Principal Investigator — NHS Lothian

REFERENCES:
- [Background] Gautherie M. Temperature and blood flow patterns in breast cancer during natural evolution and following radiotherapy. Prog Clin Biol Res. 1982;107:21-64. No abstract available. PMID 7167480
- [Background] Gautherie M, Gros CM. Breast thermography and cancer risk prediction. Cancer. 1980 Jan 1;45(1):51-6. doi: 10.1002/1097-0142(19800101)45:13.0.co;2-l. PMID 7351006
- [Background] Yahara T, Koga T, Yoshida S, Nakagawa S, Deguchi H, Shirouzu K. Relationship between microvessel density and thermographic hot areas in breast cancer. Surg Today. 2003;33(4):243-8. doi: 10.1007/s005950300055. PMID 12707816
- [Background] Barrett AH, Myers PC. Subcutaneous temperatures: a method of noninvasive sensing. Science. 1975 Nov 14;190(4215):669-71. doi: 10.1126/science.1188361.
- [Background] Tahir H, Shah E, Siores C, Daskalakis. Non-invasive devices for early detection of breast tissue oncological abnormalities using microwave radio thermometry. HalaGali-Muhtasib. Advances in Cancer Therapy. InTech, 2011; 447-476.
- [Background] Toutouzas K, Grassos C, Drakopoulou M, Synetos A, Tsiamis E, Aggeli C, Stathogiannis K, Klettas D, Kavantzas N, Agrogiannis G, Patsouris E, Klonaris C, Liasis N, Tousoulis D, Siores E, Stefanadis C. First in vivo application of microwave radiometry in human carotids: a new noninvasive method for detection of local inflammatory activation. J Am Coll Cardiol. 2012 May 1;59(18):1645-53. doi: 10.1016/j.jacc.2012.01.033. PMID 22538335
- [Background] Toutouzas K, Synetos A, Nikolaou C, Stathogiannis K, Tsiamis E, Stefanadis C. Microwave radiometry: a new non-invasive method for the detection of vulnerable plaque. Cardiovasc Diagn Ther. 2012 Dec;2(4):290-7. doi: 10.3978/j.issn.2223-3652.2012.10.09. PMID 24282729
- [Background] Klemetsen O, Birkelund Y, Jacobsen SK, Maccarini PF, Stauffer PR. DESIGN OF MEDICAL RADIOMETER FRONT-END FOR IMPROVED PERFORMANCE. Prog Electromagn Res B Pier B. 2011;27:289-306. doi: 10.2528/pierb10101204. PMID 21779411
- [Background] Bardati F, Iudicello S. Modeling the visibility of breast malignancy by a microwave radiometer. IEEE Trans Biomed Eng. 2008 Jan;55(1):214-21. doi: 10.1109/TBME.2007.899354. PMID 18232364
- [Background] Vesnin SG, Kaplan MA, Avakjan RS. Modern microwave radiometry of breast. The tumor of women reproductive systems 2008; 3: 28 -33
- [Background] Roshkova NI, Smirnova NA, Nazarov AA. Microwave radiometry of breast and the main factors which determine its efficacy. Mammalogy 2007; 3: 21-25